CLINICAL TRIAL: NCT04001114
Title: Cigarette Smoking in Smokers With and Without a Diagnosis of Schizophrenia
Brief Title: Cigarette Smoking in Smokers With and Without Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Britta Hahn, Associate Professor, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HP-00086422
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-06

CONDITIONS: Tobacco Dependence; Schizophrenia
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia

STUDY DESIGN:
Intervention Model Description: We will compare participants with and without a diagnosis of schizophrenia. Study procedures are identical for the two groups.
Who Masked: Participant, Investigator
Masking Description: Participants compare different research cigarettes. Neither the participant nor the investigators know which cigarette is of which type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers with schizophrenia (Other): This is a diagnostic group, defined independently from this study.
  Interventions: Combination Product: Sampling Research Cigarettes
- Smokers without schizophrenia (Other): This is a diagnostic group (i.e., no diagnosis of schizophrenia), defined independently from this study.
  Interventions: Combination Product: Sampling Research Cigarettes

INTERVENTIONS:
Combination Product: Sampling Research Cigarettes — Participants sample two research cigarettes, which differ in typical tobacco smoke constituents such as tar, nicotine, carbon monoxide, etc. In the Cigarette Discrimination Session, participants sample both types of cigarettes repeatedly, guess their identity (A or B) with regard to reference cigarettes, and rate their subjective effects. In the Ad Libitum Smoking Session, participants can smoke one of these cigarette types as much or as little as they like for eight hours.

SUMMARY:
Higher rates and severity of tobacco dependence in people with schizophrenia, as compared with the general population, contribute to the lower life expectancy seen in this population. Dependent tobacco smoking is controlled by how different aspects of cigarette smoking are perceived. There is evidence suggesting that people with schizophrenia differ in how they perceive cigarette smoking, which, if confirmed, would have implications for tailoring treatment interventions for smoking cessation in schizophrenia.

DETAILED DESCRIPTION:
The aim of the present study is to determine whether tobacco smoking in people with schizophrenia is governed by different aspects and effects of cigarette consumption. Smokers participating in this study either have no psychiatric diagnosis, or a diagnosis of schizophrenia or schizoaffective disorder. Over four study visits, participants will sample and compare different research cigarettes, complete questionnaires and concentration tasks, and smoke one type of research cigarette for eight hours while wearing a nicotine patch. By shaping our understanding of tobacco dependence in schizophrenia, the present project may redirect treatment development toward strategies tailored to the specific vulnerabilities of this population, which is among the most severely affected by its detrimental impact on health and life.

ELIGIBILITY:
Inclusion Criteria:

* Regular smoker of at least 10 cigarettes or cigarillos/day for at least 2 years
* For participants with schizophrenia: DSM-5 diagnosis of schizophrenia or schizoaffective disorder
* For participants with schizophrenia: Able to give informed consent
* For smokers with schizophrenia: No change in psychiatric medication or dosage in the last 4 weeks

Exclusion Criteria:

* Uncontrolled hypertension (resting systolic BP above 150 or diastolic above 95 mm Hg)
* Cardiovascular disease, such as history of myocardial infarction and ischemia, heart failure, angina, severe arrhythmias, or EKG abnormalities
* Severe asthma
* Chronic obstructive pulmonary disease
* Neurological illness, such as stroke, seizure disorder, neurodegenerative disease, or organic brain syndrome
* Mental retardation
* Alcohol or substance use disorder except nicotine within the last year
* Use of benztropine (Cogentin), varenicline (Chantix), bupropion (Wellbutrin, Zyban), or any type of nicotine replacement
* Pregnant or lactating
* For healthy control smokers: DSM-5 diagnosis of depression, bipolar disorder, ADHD, autism spectrum disorder, anorexia, bulimia nervosa, or any schizophrenia-spectrum disorder
* For healthy control smokers: immediate family history of psychosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britta Hahn, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smokers With Schizophrenia | Smokers Without Schizophrenia
Started | 18 | 13
Completed | 17 | 9
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smokers With Schizophrenia | Smokers Without Schizophrenia | Total
Number analyzed (Participants) | 18 | 13 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (11.9) | 48.3 (7.5) | 43.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 11 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 6 | 2 | 8
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 13 | 31

OUTCOME MEASURES:

1. Primary Outcome: End-of-session Carbon Monoxide
Description: The concentration (ppm) of carbon monoxide (CO) in breath is measured by exhalation into a CO breathalyzer at the end of the 8-hour Ad Libitum Smoking Session. Only very-low-nicotine-content (virtually nicotine-free) cigarettes were consumed in this session.
Time Frame: One day (in the Ad Libitum Smoking Session), over an 8-hour time frame.
Population: One smoker with schizophrenia and one smoker without schizophrenia did not complete the study session in which this measurement was obtained but completed all other study sessions.
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | Smokers With Schizophrenia | Smokers Without Schizophrenia
Number analyzed (Participants) | 16 | 8
parts per million (ppm) | 62.7 (41.7) | 43.0 (23.3)

2. Primary Outcome: Cigarette Discrimination Accuracy
Description: Participants sample 4 cigarettes of type A and 4 cigarettes of type B in a double-blind manner and indicate for each cigarette if they think it is of type A or B. Two reference trials with cigarette type unblinded will be performed before the first and fifth sample cigarette. For each sampled cigarette, the score is either 1 (correct) or 0 (incorrect). Discrimination accuracy is calculated by averaging the eight scores for each participant.
Time Frame: One day (in the Cigarette Discrimination Session), over a 6-hour time frame.
Population: One smoker with schizophrenia did not complete the study session in which this measurement was obtained, but completed the rest of the study.
Measure: Mean (Standard Deviation); unit: percentage of choices that were correct
Arm/Group | Smokers With Schizophrenia | Smokers Without Schizophrenia
Number analyzed (Participants) | 16 | 9
percentage of choices that were correct | 65.6 (31.8) | 81.9 (11.0)

3. Secondary Outcome: Change in the Number of Research Cigarettes Smoked
Description: In the Ad Libitum Smoking Session, participants can smoke as many research cigarettes (all very-low-nicotine-content) as they wish. The propensity to maintain smoking despite the absence of nicotine was quantified by subtracting the number of cigarettes smoked in the last two hours from that in the first two hours of the session. Smaller difference values indicate that smoking was upheld by very-low-nicotine-content cigarettes.
Time Frame: One day (in the Ad Libitum Smoking Session), over an 8-hour time frame.
Population: One smoker with schizophrenia and one smoker without schizophrenia did not complete the study session in which this measurement was obtained but completed the rest of the study.
Measure: Mean (Standard Deviation); unit: difference in cigarettes smoked
Arm/Group | Smokers With Schizophrenia | Smokers Without Schizophrenia
Number analyzed (Participants) | 16 | 8
difference in cigarettes smoked | 1.75 (4.30) | 1.50 (0.93)

4. Secondary Outcome: Difference in Subjective State Composite Score
Description: The measure is derived by transforming scores on the Minnesota Nicotine Withdrawal Scale (where higher values signify more withdrawal), the Affect-based Withdrawal Scale (higher values signify a worse emotional state), Questionnaire for Smoking Urges (higher values indicate more craving), and modified Cigarette Evaluation Questionnaire (mCEQ, higher values indicate greater subjective effects of smoking on mood, hunger, physiology) into standard z-scores, thus giving each scale a mean of 0 and standard deviation of 1. Withdrawal and craving scores were re-poled (inversing the sign), and scales were averaged for each subject. The resulting composite quantified the subjective state response to cigarette smoking, larger values indicating less withdrawal, less craving, and larger effects on the mCEQ. The difference therein between the research cigarettes containing nicotine and those containing almost no nicotine quantified the subjective state response to nicotine.
Time Frame: One day (in the Cigarette Discrimination Session), over a 6-hour time frame.
Population: One smoker with schizophrenia and one smoker without schizophrenia did not complete the study session in which this measurement was obtained. One additional smoker with schizophrenia did not complete the subjective state measurements but completed all other aspects of the session.
Measure: Mean (Standard Deviation); unit: difference in z-score
Arm/Group | Smokers With Schizophrenia | Smokers Without Schizophrenia
Number analyzed (Participants) | 15 | 9
difference in z-score | 0.13 (0.26) | 0.039 (0.15)

ADVERSE EVENTS:
Time Frame: There were three study days, plus the screening session, for a total of 4 days.
Arm/Group | Smokers With Schizophrenia | Smokers Without Schizophrenia
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/13
Other Adverse Events (participants affected / at risk) | 0/18 | 0/13

LIMITATIONS AND CAVEATS:
The targeted enrollment was not achieved, and sample sizes are smaller than necessary to assess all study predictions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/14/NCT04001114/Prot_SAP_000.pdf